CLINICAL TRIAL: NCT03059095
Title: Study of Yoga and Mindfulness for Psychological and Physical Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00025681
Record Dates: First submitted 2017-02-10; First posted 2017-02-23 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Psychological Trauma; PTSD
MeSH Terms: conditions — Psychological Trauma; Stress Disorders, Post-Traumatic | interventions — Yoga; Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga and Meditation (Experimental): Yoga and Meditation online sessions 2x's a week.
  Interventions: Behavioral: Yoga & Meditation

INTERVENTIONS:
Behavioral: Yoga & Meditation — Yoga is an ancient Indian science and way of life that includes the practice of specific postures, regulated breathing, and meditation.mindfulness-based stress reduction, an intervention that teaches individuals to attend to the present moment in a nonjudgmental, accepting manner

SUMMARY:
The study rationale is to analyze the extent to which adult U.S. or non U.S. veterans or active duty military personnel who participate in the Yoga for Men (YfM) online Yoga and meditation classes report changes in symptoms of psychological trauma, depression, anxiety, stress, sleep quality, and pain. The serial measurement of symptom status over a 12-month period will provide information on the trajectory of change in symptom status, as well as insight into the extent to which this program may be an effective modality for veterans and service members who are experiencing symptoms of psychological trauma, depression, anxiety, stress, sleep quality, and pain. The purpose of this study is to evaluate whether the existing YfM online program is helpful to study qualifying veterans with symptoms of PTSD and related conditions.

DETAILED DESCRIPTION:
Yoga is an ancient Indian science and way of life that includes the practice of specific postures, regulated breathing, and meditation. It is designed to bring balance and health to the physical, mental, emotional, and spiritual dimensions of the individual.

A recent systematic review of 17 studies published between the years 2011-2013 reported that most studies of yoga demonstrated positive changes in psychological or physiological outcomes related to stress. In addition, the practice of yoga also seems to be associated with moderate improvements in cognitive function , which in turn, may be expected to positively impact overall psychological well-being. These selected results provide a strong rationale to examine the effects of yoga for a range of health conditions, in addition to across various setting and by use of different delivery methods.

Much of the research on mindfulness has been in the area of anxiety and depression. Evidence suggests that mindfulness-based stress reduction, an intervention that teaches individuals to attend to the present moment in a nonjudgmental, accepting manner , can result in reduced symptoms of depression and anxiety .

ELIGIBILITY:
Inclusion/Exclusion Form

ID# __________ Visit: Screening Date: ____________________

Inclusion Criteria (all must be marked "Yes" to be eligible for the study).

1. Age 18 years or older and military service member active duty or retired Yes ___ No ___
2. Access to a computer and internet service Yes ___ No ___
3. Able to read English at 8th grade level or higher. Yes ___ No ___
4. One or more symptoms endorsed on Appendix B. Yes ___ No ___

Exclusion Criteria (must be marked "No" to be eligible for the study).

1. Never served in the military. Yes ___ No ___

Is Subject eligible for participation? Yes_____ No_____

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
PCL-5: 20 item checklist for symptoms of PTSD (PCL-5) | Accessing a change from pre, one month, six month and at one year
  There are several different ways of interpreting the scores given by the PTSD Checklist-5.[5] For a person to have a probable diagnosis of PTSD sufficient criteria must be at least moderately met in each of the four symptom groups.[1] This means you need to have one or more symptoms from questions 1 to 5, either question 6 or 7, two or more from questions 8 to 14, and two or more from questions 15 to 20, each of which must be met moderately, quite a bit or extremely.[1] In addition, a score of 38 or higher indicates probable PTSD in veterans.

SECONDARY OUTCOMES:
PSQI: 15-item Pittsburgh Sleep Quality Index (PSQI) | Accessing a change from pre, one month, six month and at one year
  measures quality and patterns of sleep in adults. It takes an estimated 3 to 6 minutes to complete. A global PSQI score greater than 5 has yielded a diagnostic sensitivity of 89.6% and specificity of 86.5% (kappa = 0.75, p<0.001) in distinguishing good and poor sleepers. Internal consistency reliability has been estimated to range from .77 to .81.

OTHER OUTCOMES:
POQ: 20-item Pain Outcomes Questionnaire (POQ) | Accessing a change from pre, one month, six month and at one year
  Short Form is a reliable and valid instrument that contains 19 primary pain items that are rated on an 11-point (0-10) Likert-type scale and one demographic question. In addition to a total pain score, six subscale scores can be calculated that correspond to: pain intensity (1 item), pain-related impairment in mobility (4 items), pain-related impairment in performing activities of daily living (4 items), sense of impairment in activity and energy levels (3 items), dysphoric affect and associated symptoms (5 items), and pain-related fear and avoidance (2 items)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: study is all online — https://yogaformen.com/pages/yoga-for-veterans